CLINICAL TRIAL: NCT02108223
Title: In This Study, the Addition of rLH, Increasing the Dose of rFSH and the Control Groups Regarding the Results of IVF in These Patients.
Brief Title: The Evaluation of Recombinant LH Supplementation in Patients With Suboptimal Response to Recombinant FSH Undergoing ICSI
Acronym: LH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Principal Investigator, fatma yazıcı yılmaz, medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4085
Record Dates: First submitted 2014-03-26; First posted 2014-04-09 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: ICSI; Suboptimal Ovarian Response; rLH
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; follitropin beta; Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fix dose r-FSH (Gonal-f) (Active Comparator): The patients who had normal ovarian response were included as the control group (Group 1). The dose of r-FSH (Gonal-f) was continued for the fix dose until the day of hCG in Group 1
  Interventions: Drug: fix dose r-FSH (Gonal-f)
- r-LH supplementation to r-FSH (Active Comparator): On day 7 of the stimulation, if at least six follicles between 6-10mm were present but there was no follicle over 10 mm on transvaginal ultrasound, E2 level was under 180 pg/ml, it has been considered that the patients had suboptimal response to the stimulation and were divided into Group 2. Group 2 received supplemental r-LH ( Lutropin alpha; Luveris, Merck Serono, France), 75IU/day to r-FSH (Gonal-f) treatment.
  Interventions: Drug: r-LH supplementation
- r-FSH (Gonal-f) (Active Comparator): Group 3: Daily 75 IU/L r-FSH was added to r-FSH treatment until the end of ovarian stimulation.
  Interventions: Drug: r-FSH (Gonal-f)

INTERVENTIONS:
Drug: fix dose r-FSH (Gonal-f) — recombinant follicle stimulation
  Other Names: puregon
  Arms: fix dose r-FSH (Gonal-f)
Drug: r-LH supplementation — recombinant luteinizing hormone
  Other Names: luveris
  Arms: r-LH supplementation to r-FSH
Drug: r-FSH (Gonal-f) — recombinant follicle stimulation hormone
  Other Names: puregon
  Arms: r-FSH (Gonal-f)

SUMMARY:
The investigators aimed to evaluate patients who had In-vitro fertilization treatment and who had COH (controlled ovarian hyperstimulation) cycles applying long protocol with GnRH (gonadotropin-releasing hormone) analogue with suboptimal response to the rFSH. The investigators evaluated and compared the addition of rLH, increasing the dose of rFSH and the control groups regarding the results of IVF in these patients.

DETAILED DESCRIPTION:
1. Aim

   -We aimed to evaluate patients who had In-vitro fertilization treatment and who had COH (controlled ovarian hyperstimulation) cycles applying long protocol with GnRH (gonadotropin-releasing hormone) analogue with suboptimal response to the rFSH. We evaluated and compared the addition of rLH, increasing the dose of rFSH and the control groups regarding the results of IVF in these patients.
2. Material and Methods -Between 01.01.2009-30.04.2011, 137 patients presented with infertility to the unit of Assisted Reproduction Techniques- of the Department of Obstetrics and Gynecology- Meram Medical Faculty- Selcuk University and were planned for ICSI-ET (intracytoplasmic sperm injection-embryo transfer) with normal ovarian function, who had long protocol of GnRH analogue and COH (controlled ovarian hyperstimulation) with rFSH were included in the study. 52 patients were considered responsive to stimulation and composed the normal control group (Group 1). On the 7th day of stimulation transvaginal ultrasonography was carried out. Patients who had at least 6 follicles about 6-10mm but had no follicle above 10mm and E2 (Oestradiol) level of <250 pg / ml were considered to have suboptimal response to stimulation and were divided into two groups. For Group 2 (n = 50), 75IU / L rLH was added to the treatment, for Group 3 (n = 35), 75IU / L of rFSH was added to the treatment. IVF results were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 23-39
* Body mass index between 18 and 30 kg/m2
* Baseline FSH ≤12 IU/l, E2 ≤ 80 pg/ml
* The presence of both ovaries and uterine cavity capable of sustaining a pregnancy
* Who had regular menstrual cycles (21-35 days) Confirmed absence of pregnancy and sufficient number of antral follicles on the transvaginal US examination on the 3rd day of menstruation
* Who were having their first or second IVF trial.

Exclusion Criteria:

* Grade III-IV endometriosis
* Clinically significant condition preventing them from undergoing gonadotrophin treatment
* More than two previous assisted cycles
* Who had a single ovary
* Unexplained gynaecological bleeding
* Polycystic ovary or an ovarian cyst of unknown aetiology
* Previously diagnosed with a space occupying lesion like submucous myoma , polyps, septum, synechia in the uterine cavity
* Have a chromosomal anomaly.

Ages: 23 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: fatma yazıcı yılmaz, MD, Principal Investigator — Sisli Etfal training and research hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fix Dose r-FSH (Gonal-f) | r-LH Supplementation to r-FSH | r-FSH (Gonal-f)
Started | 52 | 50 | 35
Completed | 52 | 50 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fix Dose r-FSH (Gonal-f) | r-LH Supplementation to r-FSH | r-FSH (Gonal-f) | Total
Number analyzed (Participants) | 52 | 50 | 35 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 50 | 35 | 137
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (3.9) | 30.3 (5.1) | 29.4 (5.1) | 29.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 35 | 137
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 52 | 50 | 35 | 137

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate
Description: percentage of participants with a pregnancy (a b-HCG determination was obtained and considered positive if the value was greater than 10 mIU/ml)
Time Frame: Up to 9 month
Population: In Group 1, transfer procedure could not be performed one patient. In Group 2, the cycle was cancelled in two patients. Oocyte could not be obtained in one patient during OPU. In other 2 patients, transfer couldn't be done. In Group 3 transfer procedure could not be performed in one patient. The pregnancy rates per embryo transfer were calculated.
Measure: Number; unit: percentage of pregnant participants
Groups:
- Fix Dose r-FSH (Gonal-f) Group 1: The patients who had normal ovarian response were included as the control group (Group 1). The dose of r-FSH (Gonal-f) was continued for the fix dose until the day of hCG in Group 1
  fix dose r-FSH (Gonal-f): recombinant follicle stimulation
- r-LH Supplementation to r-FSH Group 2: On day 7 of the stimulation, if at least six follicles between 6-10mm were present but there was no follicle over 10 mm on transvaginal ultrasound, E2 level was under 180 pg/ml, it has been considered that the patients had suboptimal response to the stimulation and were divided into Group 2. Group 2 received supplemental r-LH ( Lutropin alpha; Luveris, Merck Serono, France), 75IU/day to r-FSH (Gonal-f) treatment.
  r-LH supplementation: recombinant luteinizing hormone
- r-FSH (Gonal-f) Group 3: Group 3: Daily 75 IU/L r-FSH was added to r-FSH treatment until the end of ovarian stimulation.
  r-FSH (Gonal-f): recombinant follicle stimulation hormone
Arm/Group | Fix Dose r-FSH (Gonal-f) Group 1 | r-LH Supplementation to r-FSH Group 2 | r-FSH (Gonal-f) Group 3
Number analyzed (Participants) | 51 | 45 | 34
percentage of pregnant participants | 64.7 | 57.8 | 32.4

2. Secondary Outcome: the Number of Oocytes Retrieved
Description: median number of oocytes retrieved per participant
Time Frame: up to 9 month
Measure: Median (Standard Deviation); unit: oocytes
Arm/Group | Fix Dose r-FSH (Gonal-f) | r-LH Supplementation to r-FSH | r-FSH (Gonal-f)
Number analyzed (Participants) | 52 | 50 | 35
oocytes | 10.8 (4) | 6.6 (3.4) | 6.4 (3.3)

3. Secondary Outcome: Number of Mature Oocyte
Description: median number of mature oocytes retrieved per participant
Time Frame: up to 9 month
Measure: Median (Standard Deviation); unit: oocytes
Arm/Group | Fix Dose r-FSH (Gonal-f) | r-LH Supplementation to r-FSH | r-FSH (Gonal-f)
Number analyzed (Participants) | 52 | 50 | 35
oocytes | 8.9 (3.3) | 5.5 (2.8) | 5.5 (3)

4. Secondary Outcome: Fertilization Rate
Description: fertilization rate used to measure how many oocytes become fertilized by sperm cells
Time Frame: up to 9 month
Measure: Number; unit: percentage of fertilized oocytes
Arm/Group | Fix Dose r-FSH (Gonal-f) | r-LH Supplementation to r-FSH | r-FSH (Gonal-f)
Number analyzed (Participants) | 52 | 50 | 35
percentage of fertilized oocytes | 73.1 (20) | 74.9 (15) | 74.7 (16)

5. Secondary Outcome: Implantation Rates
Description: Implantation rate is the percentage of embryos which successfully undergo implantation
Time Frame: up to 9 months
Measure: Number; unit: percentage of embryo implantation
Arm/Group | Fix Dose r-FSH (Gonal-f) | r-LH Supplementation to r-FSH | r-FSH (Gonal-f)
Number analyzed (Participants) | 52 | 50 | 35
percentage of embryo implantation | 34.8 (15) | 36.1 (36.1) | 15 (34.7)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Fix Dose r-FSH (Gonal-f) | r-LH Supplementation to r-FSH | r-FSH (Gonal-f)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No